CLINICAL TRIAL: NCT00450489
Title: Assessment of Quality of Life and Satisfaction With Medical Care of Pediatric Type 1 Diabetes Mellitus Patients
Status: Withdrawn | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Kurt Midyett, MD, Children's Mercy Hospitals and Clinics
Other Study IDs: 07 02-030E
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2010-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Quality of Life; Satisfaction of medical care delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the change score for the PedsQL short form Diabetes and Core Modules and the Patient Assessment of Chronic Illness Care measured at baseline (before changing care delivery models) and 12 months after transitioning to the team model of care delivery.

DETAILED DESCRIPTION:
Pediatric Type 1 Diabetes Mellitus patients and their parents will complete the forms before and 12 months after the diabetes clinic at Children's Mercy Hospital in Kansas City, MO transitions to a team model of care delivery.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus six years of age and older who are receiving care in the diabetic clinic at Children's Mercy Hospital

Exclusion Criteria:

* T1 Diabetes Mellitus patients not receiving care in the diabetes clinic at Children's Mercy Hospital or not meeting the age requirements

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children cared for Type 1 Diabetes Mellitus, in Children's Mercy Hospital and Clinics, Endocrine Clinic.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Midyett, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States